CLINICAL TRIAL: NCT00810251
Title: A Multi-Site Prospective, Non-Randomized Observational Study Utilizing MatrixRIB Implants for Surgical Stabilization of Flail Chest Injuries
Brief Title: MatrixRIB Implants for Surgical Stabilization of Flail Chest Injuries: A Registry
Acronym: MatrixRIB
Status: Completed | Type: Observational
Sponsor: Legacy Biomechanics Laboratory (Other)
Collaborators: Synthes Inc. (Industry)
Responsible Party: Michael Bottlang, PhD, Director, Legacy Biomechanics Laboratory, Legacy Clinical Research & Technology Center
Other Study IDs: S08-001
Record Dates: First submitted 2008-12-16; First posted 2008-12-18 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2011-07

CONDITIONS: Flail Chest
Keywords: rib fracture; flail chest; plate; chest trauma; osteosynthesis; mechanical ventilation; respirator
MeSH Terms: conditions — Flail Chest; Rib Fractures; Thoracic Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MatrixRIB
  Interventions: Device: MatrixRIB (FDA Approval # K081623)

INTERVENTIONS:
Device: MatrixRIB (FDA Approval # K081623) — MatrixRIB implants are comprised of anatomic rib plates and intramedullary rib splints for internal surgical stabilization of rib fractures.
  Other Names: rib plates

SUMMARY:
The purpose of this observational study is to document the treatment of serial rib fractures with MatrixRIB implants in a registry.

DETAILED DESCRIPTION:
This is a multiple site, prospective, non-randomized single arm observational study. It has been designed to document the treatment of serial rib fractures with MatrixRIB implants in a registry. A flail chest is an injury in which three or more consecutive ribs are broken. This injury causes a segment of the chest wall to become unstable und prevents effective respiration. Non-operative management requires long-term mechanical ventilation and is associated with a mortality rate of 17-47%. Surgical stabilization of the rib fractures has shown to decrease this mortality by 38% - 72%. Surgical stabilization is typically performed with generic plates that require extensive bending during surgery to conform the plate to the rib in a difficult and time-consuming procedure.

The MatrixRIB system is the first implant system that has been specifically designed for fixation of flail chest injuries. It has been developed at Legacy Health System, has been extensively tested in biomechanical studies, and has been approved by the FDA. It provides anatomically contoured rib plates that can reduce the time and complexity of intra-operative plate contouring. These plates will be used in the present study in place of generic plates. It furthermore provides intramedullary rib splints that enable less invasive fixation of posterior rib fractures that are difficult to access for plate fixation.

The primary objective of this study is to document stabilization of flail chest injuries with MatrixRIB implants in a registry. Twenty consecutive patients with flail chest injury that receive surgical stabilization of rib fractures with MatrixRIB implants will be documented in the registry. Data collected will include baseline patient demographics, and information related to injury severity, surgical procedures, and post-operative recovery. The patients' functional outcome will be assessed up to the standard follow-up visit 3 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mono-lateral or bi-lateral flail chest injury and paradoxical motion of the chest wall, whereby a flail chest is defined by three or more consecutive ribs broken in at least two locations.
* Male and female patients, ages 21 to 80 years.
* Able and willing to obtain informed consent from patient or next of kin.
* Able and willing to adhere to 3-months follow-up visit

Exclusion Criteria:

* Pregnant women
* Patients who are enrolled in another investigational treatment trial.
* Severe closed head injury (AIS head > 3)
* Severe spinal injury with neurological deficit above thoraco-lumbar junction.
* Chronic preexisting heart, pulmonary, hepatic, and/or renal disease.
* Patients who are not expected to survive the follow-up period.
* Patient with an acutely paralyzed hemidiaphragm.
* Considered an inappropriate participant by the study physician.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Flail chest patients admitted to Level I and Level II trauma centers.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2008-12; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Durable flail chest stabilization, resulting in effective chest wall function at three months post surgery. | 3 months post surgery

SECONDARY OUTCOMES:
Length of ICU stay and hospitalization. | up to 3 months
Incidence of pneumonia, localized infection. | up to 3 months
Duration of post-operative requirement for ventilatory support | up to 3 months
Duration of post-operative medication for chest pain | up to 3 months
RAND 36-Item Short Form Health Survey (SF-36) | 3 months post surgery
Intra-operative complications related to fixation hardware. | intra-operative

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bottlang, PhD, Principal Investigator — Legacy Clinical Research & Technology Center
Locations (1):
- Legacy Emanuel Hospital, Portland, Oregon, United States